CLINICAL TRIAL: NCT06927752
Title: Retrospective Data Analysis PelviGYNious/EndoGYNious (PMCF-4.2-004)
Brief Title: Retrospective Data Analysis PelviGYNious/EndoGYNious
Status: Active, not recruiting | Type: Observational
Sponsor: A.M.I. Agency for Medical Innovations GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: PMCF-4.2-004
Record Dates: First submitted 2025-03-27; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Prolapse; Sacrocolpopexy; Pelvic Organ Prolapse (POP)
Keywords: Sacrocolpopexy; Sacrocervicopexy; surgical mesh; laparoscopic mesh
MeSH Terms: conditions — Prolapse; Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- EndoGYNious: Patient received EndoGYNious mesh implant.
  Interventions: Device: EndoGYNious
- PelviGYNious: Patient received PelviGYNious mesh implant.
  Interventions: Device: PelviGYNious

INTERVENTIONS:
Device: PelviGYNious — Patient received PelviGYNious implant.
  Groups: PelviGYNious
Device: EndoGYNious — Patient received EndoGYNious implant.
  Groups: EndoGYNious

SUMMARY:
The retrospective patient chart review aims to generate additional data to substantiate the safety and performance of EndoGYNious and PelviGYNious.

ELIGIBILITY:
Inclusion Criteria:

* Surgery for POP
* Implantation of either EndoGYNious or PelviGYNious
* Concomitant procedures are allowed
* Women minimum 18 years old
* Written informed consent for surgery

Exclusion Criteria:

Patients who rule out subsequent contact by the hospital will be excluded.

The use of the products is contraindicated in case of:

* pregnancy and/or patients who consider future pregnancies
* adolescent/ pubescent patients
* existence of a known sensitivity/ allergy against plastic materials such as polypropylene, polyester, etc.
* any pathology, including known or suspected uterine pathology, which would compromise placement of the implant/mesh (e.g. anatomical distortion or abnormalities)
* known anticoagulation disorder
* anticoagulant therapy
* autoimmune connective tissue disease
* renal insufficiency and upper urinary tract obstruction
* cancer illnesses of the vagina / cervix / rectum
* undergone radiation therapy on the vagina, cervix, rectum
* planned or emergency opening of the gastro-intestinal tract, as this could cause a risk of product contamination that could lead to infection that would require removal of the implant/device
* active or latent infection especially of the genital system and/or urinary tract

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The planned clinical investigation is a retrospective chart review of clinical data.
  All patients who underwent surgery between January 2016 and December 2023 and met the inclusion criteria and no exclusion criteria were analyzed.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Patient subjective outcome | From baseline to the end of last follow-up [3 months, 12 months]
  Patient subjective outcome after POP treatment with EndoGYNious or PelviGYNious will be measured with a validated questionnaire (German Pelvic Floor Questionnaire "Deutscher Beckenboden-Fragebogen") . This questionnaire focus on 4 items (bladder, bowel, prolapse, sexuality).
  Each item has its scores, scores were summed up for each category (bladder max. 45, bowel max. 34, prolapse max. 15, sexual max. 21), Calculation: (achieved value of category/ max. value of category)*10; max. value 10 for each category, max. final score 40 The postoperative scores will be compared with the preoperative scores.

SECONDARY OUTCOMES:
Postoperative complications | From baseline to the end of last follow-up [average of minimum 3 months]
  To analyze postoperative complications in women undergoing POP treatment with EndoGYNious or PelviGYNious during the follow up period. The occurrence of each complicaiton/adverse event will be compared to the occurrence of the same complication by similar products or other state of the art treatments
Anatomical success (POP-Q) | From baseline to the end of last follow-up [average of minimum 3 months]
  POP-Q system according to ICS with POP-Q stages 0, I, II, III, IV The postoperative POP-Q stages (overall, apical compartment, anterior compartment, posterior compartment) will be compared to the preoperative POP-Q stages.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Erlangen, Frauenklinik, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: No